CLINICAL TRIAL: NCT03645265
Title: Rhythmic Entrainment in Bilingual Speakers With Dysarthria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results showing no effect
Sponsor: Herbert H. Lehman College, City University of New York (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0851
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease; Ataxia
Keywords: speech rhythm; speech therapy
MeSH Terms: conditions — Parkinson Disease; Ataxia; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Single case experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gestures (Experimental): Use of hand gestures to improve speech rhythm and speech production
  Interventions: Behavioral: Gestures
- Auditory (Experimental): Use of auditory cues to improve speech rhythm and speech production
  Interventions: Behavioral: Auditory

INTERVENTIONS:
Behavioral: Auditory — Use of auditory cues to improve speech production
  Arms: Auditory
Behavioral: Gestures — Use of gestures to improve speech production
  Arms: Gestures

SUMMARY:
The objectives of this study are to determine i) the effect of rhythmic entrainment of speech with hand gestures and auditory rhythmic cues on intelligibility and speech naturalness in Spanish-accented speakers of English in two pathology groups: ataxic dysarthria and hypokinetic dysarthria secondary to idiopathic Parkinson's disease; and ii) the extent to which speech rate and effort are control parameters of entrainment. These objectives will be achieved with the following specific aims:

Specific Aim 1: Determine the effect of three rates of hand gestures and auditory rhythmic cues and the degree to which learning and carry-over occur.

Specific Aim 2: Determine the effect of increased speech effort, operationalized as clear speech, and the interaction effect of clear speech with hand gestures and auditory rhythmic cues.

Specific Aim 3: Investigate the perception of speech rhythm and its relationship to entrainment.

DETAILED DESCRIPTION:
The objectives of this study are to determine i) the effect of rhythmic entrainment of speech with hand gestures and auditory rhythmic cues on intelligibility and speech naturalness in Spanish-accented speakers of English in two pathology groups: ataxic dysarthria and hypokinetic dysarthria secondary to idiopathic Parkinson's disease; and ii) the extent to which speech rate and effort are control parameters of entrainment. These objectives will be achieved with the following specific aims:

Specific Aim 1: Determine the effect of three rates of hand gestures and auditory rhythmic cues and the degree to which learning and carry-over occur.

Specific Aim 2: Determine the effect of increased speech effort, operationalized as clear speech, and the interaction effect of clear speech with hand gestures and auditory rhythmic cues.

Specific Aim 3: Investigate the perception of speech rhythm and its relationship to entrainment.

The protocol calls for 12 talkers to participate in a single case experimental design: 6 Spanish-accented speakers of English and 6 native English speakers, and each language group consisting of 2 healthy controls, 2 adults diagnosed with ataxic dysarthria and 2 adults diagnosed with hypokinetic dysarthria secondary to idiopathic Parkinson's disease. Sixty monolingual healthy adult listeners will rate intelligibility, accentedness, and ease of understanding.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease (4) or dysarthria secondary to ataxia (4) or healthy (4)
* monolingual speaker of American English (6) or native speaker of Spanish who speaks English with a Spanish accent (6)
* age 21 or older

Exclusion Criteria:

* Cognitive impairment that prevents participation in the therapy
* Fluent speakers of languages other than English or Spanish
* younger than 21 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Intelligibility | immediately upon completion of the therapy
  Intelligibility = the accuracy with which a listener understands a speaker. It will be measured by having the subjects undergoing the therapy ("the talkers") read 28 phrases using accompanying gesture or auditory cues and listeners will transcribe the sentences. The number of words accurately transcribed / the number of words in the phrase = intelligibility score for each phrase per listener

SECONDARY OUTCOMES:
Ease of understanding | Immediately upon completion of the therapy
  Ease of understanding = the ease with which listeners understand the speakers. It will be measured by having the subjects undergoing the therapy ("the talkers") read 28 phrases using accompanying gesture or auditory cues and listeners will rate how easy it is to understand the talkers using a 0 to 9 visual analog scale with 0 = very easy and 9= very hard, for each phrase per listener
Speech naturalness | immediately upon completion of the therapy
  Speech naturalness = the degree to which the listeners consider the speakers to have natural or unnatural speech. It will be measured by having the subjects undergoing the therapy ("the talkers") read 28 phrases using accompanying gesture or auditory cues and listeners will rate how natural-sounding the talker sounds by using a 0 to 9 visual analog scale with 0 = very natural and 9 = very unnatural, for each phrase per listener

CONTACTS AND LOCATIONS:
Overall Officials: Alison Behrman, PhD, Principal Investigator — Lehman College
Locations (1):
- Lehman College, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study and publication of the data
Access Criteria: Researchers who have contacted me directly with clear purpose and plan for use of data and then have IRB approval.